CLINICAL TRIAL: NCT01751321
Title: Glucose Variability With DPP-4 Inhibition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Research Clinical Centre of the Russian Railways, JSC (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40591
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- sitagliptin, metformin, placebo (Other): 1. group- 25 patients will take sitagliptin 50 mg and metformin 1000 mg twice in a day
  2. group- 25 patients will take placebo 50 mg and metformin 1000 mg twice in a day
  Interventions: Drug: Sitagliptin, placebo

INTERVENTIONS:
Drug: Sitagliptin, placebo — sitagliptin 50 / metformin 1000 twice in a day and placebo 50 mg /metformin 1000 twice in a day
  Other Names: Januvia

SUMMARY:
Glucose Variability With DPP-4 Inhibition

DETAILED DESCRIPTION:
Patients with Type 2 Diabetes, age 35-75y., will be included in this double blind randomized placebo controlled study.

The sample size of 50 patients completing the 30 day study period is based on statistical input from Merck Research Laboratories, Rahway NJ.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* receiving a stable dose of metformin ≥ 1500 mg
* HbA1c 7,5% -10/0 %

Exclusion Criteria:

* Type 1 diabetes
* HbA1c < 7,5% and > 10,0%

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
glucose variability | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ametov, MD, Principal Investigator — Research Clinical Centre of the Russian Railways, JSC